CLINICAL TRIAL: NCT04682886
Title: Research on Key Techniques for Intelligent Diagnosis and Ablation Decision-making of Liver Cancer and Evolution by Contrast-enhanced Ultrasound
Brief Title: Radiomics Analysis of Focal Liver Lesions Based on Contrast-Enhanced Ultrasound Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ping Liang (Other)
Responsible Party: Sponsor-Investigator, Ping Liang, Prof, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: 82030047
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Focal Liver Lesions; Contrast-enhanced Ultrasound
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: diagnosis — there is no intervention diagnosis or treatment for patients

SUMMARY:
Contrast-enhanced ultrasound (CEUS) substantially improves the potential of ultrasound (US) for the identification and characterization of focal liver lesions (FLLs). Compared to contrasted-enhanced MRI and CT, it has some unique advantages, such as the absence of ionizing radiation, and easy operability and repeatability. However, the efficacy of CEUS in diagnosing liver lesions is challenged by several factors including being highly dependent on doctor's experience, low signal-to-noise ratio, and low interobserver agreement. Therefore, it is a beneficial attempt to construct an intelligent CEUS diagnosis system using digital information technology. This study aims to collect standard data of CEUS cines recordings and develop deep learning model for accurate segmentation, detection and classification of liver lesions.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a solid liver tumor visible during routine ultrasound and received CEUS.
2. disease history and standard of reference of the lesions can be acquired

Exclusion Criteria:

1. hypersensitivity for ultrasound contrast media
2. pregnant or lactating patients
3. previously treated lesions or local relapse from previously treated lesions
4. diffuse tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with focal liver lesions
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC value | through study completion, an average of 7 year
  Area under the receiver operating characteristic (ROC) curve (AUC）
specificity | through study completion, an average of 7 year
  diagnosis specificity of intelligent CEUS analysis
sensitivity | through study completion, an average of 3 year
  diagnosis sensitivity of intelligent ultrasound analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ding W, Li B, Zhao L, Zheng L, Li X, Liu S, Yu J, Liang P. Improving Detection of Intrahepatic Cholangiocarcinoma with a Contrast-enhanced US-based Deep Learning Model. Radiol Imaging Cancer. 2025 Nov;7(6):e250078. doi: 10.1148/rycan.250078. PMID 41236388
- [Derived] Wu J, Liu S, Zhang Y, Ding W, Zhao Q, Wang Y, Xiao F, Yu X, Xie X, Liu S, Zhao J, Liao J, Yu J, Liang P. Prediction of Macrotrabecular-Massive Hepatocellular Carcinoma and Associated Prognosis Using Contrast-enhanced US and Clinical Features. Radiol Imaging Cancer. 2025 Jul;7(4):e240419. doi: 10.1148/rycan.240419. PMID 40607931
- [Derived] Ding W, Meng Y, Ma J, Pang C, Wu J, Tian J, Yu J, Liang P, Wang K. Contrast-enhanced ultrasound-based AI model for multi-classification of focal liver lesions. J Hepatol. 2025 Aug;83(2):426-439. doi: 10.1016/j.jhep.2025.01.011. Epub 2025 Jan 21. PMID 39848548